CLINICAL TRIAL: NCT01133665
Title: Phase II Study of Cetuximab and Lenalidomide in Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Cetuximab and Lenalidomide in Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-206-B
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Squamous Cell Carcinoma
Keywords: Head and Neck, Squamous Cell; Recurrent or metastatic squamous cell or undifferentiated carcinoma of the head and neck that is not amenable to curative therapy
MeSH Terms: conditions — Carcinoma, Squamous Cell; Recurrence | interventions — Cetuximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sub Group 1 (Experimental): All Subjects Enrolled in the Trial
  Interventions: Drug: Cetuximab and Lenalidomide

INTERVENTIONS:
Drug: Cetuximab and Lenalidomide — The treatment of Head and Neck Cancer with Cetuximab and Lenalidomide

SUMMARY:
The purpose of this study is to study specific FcRIIIa polymorphisms and their correlation with clinical outcome in subjects treated with cetuximab and lenalidomide.

DETAILED DESCRIPTION:
To study specific FcRIIIa polymorphisms and their correlation with clinical outcome in subjects treated with cetuximab and lenalidomide. There is evidence with cetuximab in CRC, trastuzumab in breast cancer and rituximab with follicular lymphoma, that FcRIIIa polymorphisms correlate with clinical response to antibody therapy and clinical outcome. It is our hypothesis that patients with SCCHN will have clinical outcomes to cetuximab and lenalidomide that correlate with patient FcRIIIa genotype.

Secondary:

To evaluate the safety and toxicity profile of the combination of cetuximab and lenalidomide given to treat subjects with SCCHN.

To study FcRIIIa polymorphisms and the correlation with the ability of NK cells to mediate ADCC against SCCHN. It is our hypothesis that NK cells from patients with advanced SCCHN can mediate ADCC against SCCHN cell lines in the presence of cetuximab and lenalidomide and that the efficiency of ADCC correlates with FcRIIIa polymorphisms.

To evaluate the ability of NK cells to induce ADCC expression of specific activation markers on the NK cell surface. It is our hypothesis that NK cells that induce ADCC will express specific activation markers that are predictive of efficiency of ADCC.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age ≥18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Recurrent or metastatic squamous cell or undifferentiated carcinoma of the head and neck that is not amenable to curative therapy. Patients who are candidates for local or locoregional therapy should not be deprived of proven beneficial palliative therapies.
5. All previous cancer therapy, including radiation, hormonal therapy, EGFR inhibitors, and surgery, must have been discontinued at least 4 weeks prior to treatment in this study.
6. ECOG performance status of 0-1 at study entry.
7. Laboratory test results within these ranges:

   * Absolute neutrophil count to ≥ 1000/mm³
   * Platelet count ≥ 100,000/mm³
   * Calculated creatinine clearance ≥ 50ml/min by Cockcroft-Gault estimation
   * Total bilirubin < 1.5 x ULN
   * AST (SGOT) and ALT (SGPT) < 3 x ULN or < 5 x ULN if hepatic metastases are present.
8. Disease free of prior malignancies for < 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in-situ" of the cervix or breast. Patients with malignancies diagnosed less than 3 years prior to study entry are eligible if the first cancer was no greater than stage I and did not recur. Patients with malignancies diagnosed less than 3 years prior to study entry must have the diagnosis of recurrent or metastatic squamous cell carcinoma of the head and neck confirmed pathologically.
9. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
10. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
11. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
12. Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded), with minimum lesion size ≥ 2 cm on conventional measurement techniques or ≥ 1 cm on spiral computed tomography (CT) scan. Lesions that can be measured clinically must be at least 1 cm in greatest dimension by caliper measurement.

Exclusion Criteria:

1. Primary head and neck carcinomas of the salivary gland, skin, or thyroid regardless of pathology
2. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
3. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
4. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
5. Use of any other experimental drug or therapy within 28 days of baseline.
6. Prior therapy with lenalidomide for squamous cell carcinoma of the head and neck
7. Known hypersensitivity to thalidomide.
8. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
9. Concurrent use of other anti-cancer agents or treatments.
10. Known positive for HIV or infectious hepatitis, type B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, M.D., Study Chair — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- See also: The University of Chicago Cancer Research Center Website — http://uccrc.uchicago.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetuximab and Lenalidomide: Patients with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) were treated wıth cetuximab (500 mg/m2 IV every 2 weeks) and lenalidomide (25 mg orally or via feeding tube once daily)
Period: Overall Study
Arm/Group | Cetuximab and Lenalidomide
Started | 42
Completed | 40
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 59 [42 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Correlate the Presence of Specific Fc RIIIa Polymorphisms With Progression-free Survival in Subjects Receiving Cetuximab and Lenalidomide for SCCHN.
Description: Progression-free survival (PFS) was defined as time from date of the first treatment dose administered to the earlier of disease progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 24 months
Measure: Median (Full Range); unit: months
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
months | 1.8 [1.0 to 11.7]

2. Secondary Outcome: Number of Participants With Fatigue Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: The number of participants for analysis was determined with >5% incidence of adverse events or any grade 3-4 adverse events related to cetuximab/lenalidomide
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 33
  Grade 3-4 | 2

3. Secondary Outcome: Number of Participants With Maculopapular Rash Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 27
  Grade 3-4 | 0

4. Secondary Outcome: Number of Participants With Constipation Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 16
  Grade 3-4 | 0

5. Secondary Outcome: Number of Participants With Anemia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 14
  Grade 3-4 | 3

6. Secondary Outcome: Number of Participants With Anorexia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 12
  Grade 3-4 | 1

7. Secondary Outcome: Number of Participants With Nausea Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 10
  Grade 3-4 | 0

8. Secondary Outcome: Number of Participants With Hypoalbuminemia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 9
  Grade 3-4 | 0

9. Secondary Outcome: Number of Participants With Lymphopenia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 9
  Grade 3-4 | 7

10. Secondary Outcome: Number of Participants With Oral Mucositis Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 9
  Grade 3-4 | 0

11. Secondary Outcome: Number of Participants With Pain Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 8
  Grade 3-4 | 0

12. Secondary Outcome: Number of Participants With Vomiting Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 8
  Grade 3-4 | 0

13. Secondary Outcome: Number of Participants With White Blood Cell Decreased Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 8
  Grade 3-4 | 5

14. Secondary Outcome: Number of Participants With Diarrhea Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 7
  Grade 3-4 | 1

15. Secondary Outcome: Number of Participants With Hyponatremia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 7
  Grade 3-4 | 3

16. Secondary Outcome: Number of Participants With Neutropenia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 7
  Grade 3-4 | 6

17. Secondary Outcome: Number of Participants With Headache Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 6
  Grade 3-4 | 1

18. Secondary Outcome: Number of Participants With Hypokalemia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 6
  Grade 3-4 | 1

19. Secondary Outcome: Number of Participants With Hypophosphatemia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 6
  Grade 3-4 | 1

20. Secondary Outcome: Number of Participants With Thrombocytopenia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 6
  Grade 3-4 | 4

21. Secondary Outcome: Number of Participants With Acneiform Rash Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 6
  Grade 3-4 | 0

22. Secondary Outcome: Number of Participants With Hyperglycemia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 5
  Grade 3-4 | 0

23. Secondary Outcome: Number of Participants With Alkaline Phosphatase Increased Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 4
  Grade 3-4 | 0

24. Secondary Outcome: Number of Participants With Aspartate Aminotransferase Increased Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 4
  Grade 3-4 | 0

25. Secondary Outcome: Number of Participants With Xerostomia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 3
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 6
  Grade 3-4 | 0

26. Secondary Outcome: Number of Participants With Fever Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 4
  Grade 3-4 | 0

27. Secondary Outcome: Number of Participants With Hypocalcaemia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 4
  Grade 3-4 | 0

28. Secondary Outcome: Number of Participants With Neck Pain Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 4
  Grade 3-4 | 0

29. Secondary Outcome: Number of Participants With Peripheral Sensory Neuropathy Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: Analysis Population Description: The number of participants for analysis was determined with >5% incidence of adverse events or any grade 3-4 adverse events related to cetuximab/lenalidomide
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 4
  Grade 3-4 | 0

30. Secondary Outcome: Number of Participants With Alanine Aminotransferase Increased Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 3
  Grade 3-4 | 0

31. Secondary Outcome: Number of Participants With Back Pain Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 3
  Grade 3-4 | 0

32. Secondary Outcome: Number of Participants With Dyspnea Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 3
  Grade 3-4 | 0

33. Secondary Outcome: Number of Participants With Weight Loss Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 3
  Grade 3-4 | 0

34. Secondary Outcome: Number of Participants With Blood Bilirubin Increased Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 2
  Grade 3-4 | 1

35. Secondary Outcome: Number of Participants With Infusion Related Reaction Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 2
  Grade 3-4 | 1

36. Secondary Outcome: Number of Participants With C. Diff Infection Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 1
  Grade 3-4 | 1

37. Secondary Outcome: Number of Participants With Febrile Neutropenia Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 1
  Grade 3-4 | 1

38. Secondary Outcome: Number of Participants With Lymphocyte Count Increased Related to Cetuximab/Lenalidomide
Description: Toxicity was scored according to NCI/CTC version 4
Time Frame: 24 month
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Cetuximab and Lenalidomide
Number analyzed (Participants) | 40
participants
  All grades | 1
  Grade 3-4 | 1

ADVERSE EVENTS:
Arm/Group | Cetuximab and Lenalidomide
Serious Adverse Events (participants affected / at risk) | 16/40
Other Adverse Events (participants affected / at risk) | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab and Lenalidomide (N=40)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Death (General disorders) | 3
Fever (General disorders) | 3
Infusion related reaction (General disorders) | 1
Skin infection (Infections and infestations) | 1
INR increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab and Lenalidomide (N=40)
Anemia (Blood and lymphatic system disorders) | 15
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 17
Diarrhea (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 6
Mucositis oral (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 11
Oral pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 8
Facial pain (General disorders) | 3
Fatigue (General disorders) | 33
Fever (General disorders) | 6
Pain (General disorders) | 8
Papulopustular rash (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 9
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 6
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 12
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes